CLINICAL TRIAL: NCT06303206
Title: Telehealth for Emergency-Community Continuity of Care Connectivity Via Home Telemonitoring for Blood Pressure Randomized Controlled Trial
Brief Title: TEC4Home Blood Pressure Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Karen Tran, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H23-00623
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Blood Pressure Telemonitoring (HBPT) + Case Management (CM) (Experimental): This group will be asked to follow home BP monitoring as per instructions. Results will be transmitted and telemonitored using an app, where case managers (designated pharmacists) will monitor BP values to provide counselling for medication adherence and behavioural support and review telemonitored BP summaries and adjust BP medications according to protocol. Case management teams will contact participants at baseline and every month until the end of the study, or more frequently if BP is uncontrolled.
  Interventions: Device: Home Blood Pressure Telemonitoring (HBPT) + Case Management (CM)
- Usual Care (No Intervention): This group will receive usual care by their primary care provider and provided with hypertension education materials similar to the intervention group. Participants will receive the same home BP monitor to encourage monitoring of home BP based on hypertension guideline recommendations. Home BP readings will tele-transmit via the app for study purposes, but not made available to the case managers or primary care providers, except if necessary for safety reasons, or at the discretion of the data safety monitoring physician.

INTERVENTIONS:
Device: Home Blood Pressure Telemonitoring (HBPT) + Case Management (CM) — Home Blood Pressure Telemonitoring (HBPT) includes used of an app to collect and transmit blood pressure readings.
  Case Management (CM) includes pharmacists reviewing BP data and providing counselling to participants based on their BP values.
  Arms: Home Blood Pressure Telemonitoring (HBPT) + Case Management (CM)

SUMMARY:
The goal of this clinical trial is to evaluate the effect of home blood pressure telemonitoring (HBPT) and case management (CM), relative to usual care, for improving blood pressure (BP) control among patients with high blood pressure discharged from the emergency department (ED).

The main question it aims to answer is: Does telemonitoring with case management improve BP control, relative to usual care, for people with high blood pressure discharged from the ED?

Secondary research questions will address:

1. How do these interventions (telemonitoring and case management) improve medication adherence?
2. Do these interventions reduce physician and ED visits?
3. Are these interventions safe?
4. How do these interventions influence patient experience?

Participants in the intervention group will receive training and use of a home BP telemonitor with tele-transmission function for 12-months plus pharmacist case management to provide behavioral counseling, facilitate medication adherence, review telemonitored BP data, and adjust medications. The control group will receive usual care from their primary care physician and will receive the same home BP monitor and hypertension education.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥ 18 years of age
* Elevated triage BP AND increased average BP in three subsequent repeated measurements that are spaced at least 30 minutes after triage (systolic BP ≥ 160 mm Hg or diastolic BP ≥ 100 mm Hg)
* Own a smart phone
* Willing to measure and tele-transmit home BP readings

Exclusion Criteria:

* Hypertensive emergencies with evidence of end-organ damage, stroke, or acute coronary syndrome
* Pregnant women
* Acute intoxication
* Acute surgical or trauma patients
* Psychiatrically unstable patients
* Advanced cognitive impairment
* Patient requiring admission to hospital
* Inability to use or care for home BP monitor correctly
* From nursing home
* Unstable housing
* Non-English speaking or no family members who can help translate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure controlled | 12-months
  Comparison of proportion of participants in intervention group versus control group achieving 24h daytime SBP control (< 135 mm Hg or < 130 mm Hg if diabetic)

SECONDARY OUTCOMES:
Impact of intervention on other blood pressure measures | 6-months and 12-months
  Ambulatory BP 24h average SBP 24h average DBP 24h daytime average SBP 24h daytime DBP 24h nighttime SBP 24h nighttime DBP
  Home BP Home SBP average Home DBP average
  Proportion achieving 24h daytime DBP control (< 85 mm Hg or < 80 mm Hg if diabetic)

IPD SHARING:
Plan to Share IPD: No